CLINICAL TRIAL: NCT05872672
Title: Assessment of a Behavioral Sleep Program Using Subjective and Objective Measures of Sleep Quality in a Population With Sleep Disturbances
Brief Title: Assessment of a Behavioral Sleep Program in a Population With Sleep Disturbances
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Virginia Polytechnic Institute and State University (Other)
Responsible Party: Principal Investigator, Ulrich Kirk, Associate Professor, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 3425432
Record Dates: First submitted 2023-05-08; First posted 2023-05-24 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Sleep Disturbance
MeSH Terms: conditions — Parasomnias | interventions — Waiting Lists

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep Program (Active Comparator)
  Interventions: Behavioral: Sleep Program
- Waitlist (Other)
  Interventions: Other: Waitlist

INTERVENTIONS:
Behavioral: Sleep Program — Participants will complete the Headspace Health Sleep Program, which is an 18 day program based on CBTi, and includes the following intervention components: 1) a sleep diary to monitor sleep and associated factors; 2) cognitive interventions to address maladaptive thoughts related to sleep; 3) behavioral interventions to address maladaptive behaviors related to sleep (e.g., sleep hygiene, stimulus control, and sleep restriction); 4) de-arousal techniques (e.g., mindfulness, breathing, and muscle relaxation exercises).
  Arms: Sleep Program
Other: Waitlist — Participants will continue their regular sleep routines for an 18 day period and will not be assigned to an intervention.
  Arms: Waitlist

SUMMARY:
Sleep disturbances are considered a significant public health concern. The prevalence of disrupted sleep among US adults has increased to alarming levels. Around 70 million Americans suffer from a sleep disturbance. Reduced sleep and poor sleep quality have been linked to cardiovascular disease, increased risk for obesity, hypertension, heart attack, and stroke.

Sleep disturbances are characterized by dissatisfaction with sleep quality or sleep quantity, which may be associated with difficulties initiating sleep, difficulties maintaining sleep, or early-morning awakenings with an inability to return to sleep. Sleep disturbances including insomnia can be treated with pharmacological treatments. However, individuals often report adverse side effects. Increasing attention has therefore been paid to behavioral and psychological interventions, such as cognitive behavioral therapy and mindfulness.

The study will assess a smartphone-based sleep program by Headspace Health that combines cognitive behavioral therapy for insomnia (CBTi) and mindfulness concepts to minimize nocturnal symptoms and waking consequences associated with sleep disturbances.

The study aims to test the effectiveness of the Headspace Health Sleep Program on self-reported outcomes related to sleep quality. A secondary aim is to test objective measures of sleep quality using actigraphy.

The Headspace Health Sleep Program is an 18 day program based on CBTi, which includes the following intervention components: 1) a sleep diary to monitor sleep and associated factors; 2) cognitive interventions to address maladaptive thoughts related to sleep; 3) behavioral interventions to address maladaptive behaviors related to sleep (e.g., sleep hygiene, stimulus control, and sleep restriction); 4) de-arousal techniques (e.g., mindfulness, breathing, and muscle relaxation exercises).

DETAILED DESCRIPTION:
The purpose of the study is to examine the effectiveness of the Headspace Health Sleep Program for improving both subjective sleep quality (i.e., self-reported surveys) as well as objective sleep quality (i.e. actigraphy) in a population with sleep disturbances. The study will employ a 2-arm app-based intervention involving 1 active intervention (i.e., Headspace Health Sleep Program) and a waitlist control for a duration of 18 days.

A set of outcome measures will be used to evaluate the Headspace Health Sleep Program vs. a waitlist control group. The Insomnia Severity Index (ISI) will be used as a primary outcome measure as well as the Sleep Diary, and actigraphy. In addition, secondary outcome measures include Pittsburgh Sleep Quality Index (PSQI), Perceived Stress Scale (PSS-10), Patient Health Questionnaire-8 (PHQ-8), General Anxiety Disorder-7 (GAD-7) and Mindful Attention Awareness Scale (MAAS). Baseline measures will be taken prior to randomization, and at post-intervention. 2 weeks following the post-intervention assessment, participants will again be asked to report sleep quality using self-reported surveys.

Eligible participants will complete a 1-week baseline assessment period. Participants will be supplied with a wrist actigraph and sleep diary. On the first day of the assessment period, participants will be instructed to start wearing the wrist actigraph. They will also be instructed to complete the sleep diary the following morning. Participants will continue this procedure of filling in the sleep diary every morning for the 1-week baseline assessment period and wearing the wrist actigraph. Following the 1-week baseline assessment period, participants will be asked to return the sleep diary, wrist actigraph, and complete baseline questionnaires (i.e., ISI, PSQI, PSS-10, PHQ8, GAD7, MAAS). They will then be randomized into one of two groups (Headspace Health Sleep Program or waitlist control). Having completed the intervention, participants will be scheduled for the 1-week post-intervention assessment period. Participants will again be supplied with a wrist actigraph, and sleep diary. At the end of this 1-week post-intervention assessment period, participants will return the sleep diary, wrist actigraph, and complete questionnaires (i.e., ISI, PSQI, PSS-10, PHQ8, GAD7, MAAS). 2 weeks following the post-intervention, participants will be asked to complete the sleep diary for a 1-week follow-up assessment period and in addition the ISI, PSQI, PSS-10, PHQ8, GAD7 and MAAS.

ELIGIBILITY:
Inclusion Criteria:

* A total score of 11 or greater on the Insomnia Severity Index (ISI).
* Fluency in English
* Own a smartphone that can support downloaded apps

Exclusion Criteria:

* Completed CBTi program in the past 6 months.
* Risk factors associated with severe insomnia such as depression and self-harm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Insomnia Severity Index (ISI) | Change from baseline to immediately post-intervention and 2-week follow-up
  The ISI is a measure of sleep disturbance severity. ISI is a 7-item, self-report measure for the evaluation of insomnia. Items in the ISI concern difficulties falling asleep, problems staying asleep, daytime symptoms connected to the sleeping problem, and worrying about sleeping too little. Each item is rated from 0 to 4, giving the rating scale a maximum summed score of 28 points. According to the guidelines for interpretation, 0-7 should be interpreted as no clinically significant insomnia, 8-14 as subthreshold insomnia, 15-21 as clinical insomnia of moderate severity, and 22-28 as severe clinical insomnia.
Sleep Diary | Change from baseline to immediately post-intervention and 2-week follow-up
  Participants will be asked to complete a daily sleep diary for the duration of the 1-week baseline assessment period and the 1-week post-intervention assessment and the 1-week follow-up period. The sleep diary will be used to measure sleep efficiency (SE) and total wake time (TWT). Sleep efficiency will be calculated by dividing the amount of time sleeping in bed by the amount of time spent in bed. Total sleep time will be calculated as the total amount of nightly sleep. In addition, the sleep diary will measure sleep onset latency (SOL), wake after sleep onset (WASO). The sleep diary data will be averaged across one week with a minimum of 4 nights required for inclusion.
Actigraphy | Change from baseline to immediately post-intervention
  A wrist actigraph will be worn on the non-dominant wrist of participants for the duration of the 1-week baseline assessment period and the 1-week post-intervention assessment period. In this study the investigators will use the research-grade GT3X actigraph (wGT3X-BT: ActiGraph, Pensacola, Florida, USA), which is a small (10.5 × 30.3 × 40.6 mm) and lightweight (19 g) triaxial accelerometer and is a research-grade device. The investigators will use the ActiLife (Version 6.13.1, ActiGraph, Pensacola, Florida, USA) data analysis software to extract the variables of interest. An algorithm yields approximate values for sleep efficiency, sleep onset latency, wake after sleep onset, movement time, total wake time (TWT) and sleep fragmentation. Participants will be instructed to wear the wrist actigraph continuously in the 1-week baseline and 1-week post intervention periods. Actigraphy data will be averaged across one week with a minimum of 4 nights required for inclusion.

SECONDARY OUTCOMES:
The Pittsburgh Sleep Quality Index (PSQI) | Change from baseline to immediately post-intervention and 2-week follow-up
  The PSQI is a self-rated questionnaire which assesses sleep quality and disturbances. 19 individual items generate seven component scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The sum of scores for these seven components yields one global score. Higher scores indicate worse sleep quality where poor sleep will be a PSQI total score of > 5.
Perceived Stress Scale (PSS-10) | Change from baseline to immediately post-intervention and 2-week follow-up
  The PSS is a 10-item scale designed to measure the perception of stress within the past month. Participants use a Likert scale with responses ranging from 0 = never to 4 = very often. PSS-10 scores range from 0-40 with higher scores indicating higher perceived stress. Additionally, scores can be categorized as low (0-13), moderate (14-26), and high (27-40) perceived stress.
Patient Health Questionnaire-8 (PHQ8) | Change from baseline to immediately post-intervention and 2-week follow-up
  The PHQ-8 is used to measure depression symptoms. The PHQ-8 consists of 8 items. Participants use a Likert scale ranging from 0 = not at all to 3 = nearly every day. The range of PHQ-8 scores is 0-24.
General Anxiety Disorder-7 (GAD-7) | Change from baseline to immediately post-intervention and 2-week follow-up
  The GAD-7 is a 7-item self-report scale based on the Diagnostic and Statistical Manual of Mental Disorders-IV criteria for generalized anxiety disorder, with items scored from 0 (not at all) to 3 (nearly every day).
Mindful Attention Awareness Scale (MAAS) | Change from baseline to immediately post-intervention and 2-week follow-up
  Mindfulness will be measured by the MAAS. The MAAS is a 15-item scale designed to assess a core characteristic of dispositional mindfulness. Each of the 15 items aims at measuring one's awareness of what is taking place at the present. The MAAS is answered on a five-point Likert scale. Higher scores reflect higher dispositional mindfulness.
Sleep medication | Change from baseline to immediately post-intervention and 2-week follow-up
  Change in sleep medication will be assessed. Specifically, prescribed sleep medication, over-the-counter sleep aids, therapy, psychotropic medications (SSRIs/anxiety meds).

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Kirk, PhD, Principal Investigator — University of Southern Denmark
Locations (1):
- Fralin Biomedical Research Institute at VTC, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
Aggregated data collected in this project will be de-identified and made available on a shared secured data repository. Results from this project will be shared and disseminated, including manuscripts will be written and submitted for publication in peer-reviewed journals/conferences. All necessary ethical approvals will be obtained.
Time Frame: Data will be made available upon request after dissemination of results.

REFERENCES:
- [Background] Altman NG, Izci-Balserak B, Schopfer E, Jackson N, Rattanaumpawan P, Gehrman PR, Patel NP, Grandner MA. Sleep duration versus sleep insufficiency as predictors of cardiometabolic health outcomes. Sleep Med. 2012 Dec;13(10):1261-70. doi: 10.1016/j.sleep.2012.08.005. Epub 2012 Nov 8. PMID 23141932
- [Background] Anderson T, Corneau G, Wideman L, Eddington K, Vrshek-Schallhorn S. The impact of prior day sleep and physical activity on the cortisol awakening response. Psychoneuroendocrinology. 2021 Apr;126:105131. doi: 10.1016/j.psyneuen.2021.105131. Epub 2021 Jan 14. PMID 33493753
- [Background] Arble DM, Bass J, Behn CD, Butler MP, Challet E, Czeisler C, Depner CM, Elmquist J, Franken P, Grandner MA, Hanlon EC, Keene AC, Joyner MJ, Karatsoreos I, Kern PA, Klein S, Morris CJ, Pack AI, Panda S, Ptacek LJ, Punjabi NM, Sassone-Corsi P, Scheer FA, Saxena R, Seaquest ER, Thimgan MS, Van Cauter E, Wright KP. Impact of Sleep and Circadian Disruption on Energy Balance and Diabetes: A Summary of Workshop Discussions. Sleep. 2015 Dec 1;38(12):1849-60. doi: 10.5665/sleep.5226. PMID 26564131
- [Background] Bastien CH, Vallieres A, Morin CM. Validation of the Insomnia Severity Index as an outcome measure for insomnia research. Sleep Med. 2001 Jul;2(4):297-307. doi: 10.1016/s1389-9457(00)00065-4. PMID 11438246
- [Background] Brown KW, Ryan RM. The benefits of being present: mindfulness and its role in psychological well-being. J Pers Soc Psychol. 2003 Apr;84(4):822-48. doi: 10.1037/0022-3514.84.4.822. PMID 12703651
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Buysse DJ, Thompson W, Scott J, Franzen PL, Germain A, Hall M, Moul DE, Nofzinger EA, Kupfer DJ. Daytime symptoms in primary insomnia: a prospective analysis using ecological momentary assessment. Sleep Med. 2007 Apr;8(3):198-208. doi: 10.1016/j.sleep.2006.10.006. Epub 2007 Mar 23. PMID 17368098
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Cunnington D, Junge MF, Fernando AT. Insomnia: prevalence, consequences and effective treatment. Med J Aust. 2013 Oct 21;199(8):S36-40. doi: 10.5694/mja13.10718. PMID 24138364
- [Background] Grandner MA, Schopfer EA, Sands-Lincoln M, Jackson N, Malhotra A. Relationship between sleep duration and body mass index depends on age. Obesity (Silver Spring). 2015 Dec;23(12):2491-8. doi: 10.1002/oby.21247. Epub 2015 Nov 2. PMID 26727118
- [Background] Grandner MA, Chakravorty S, Perlis ML, Oliver L, Gurubhagavatula I. Habitual sleep duration associated with self-reported and objectively determined cardiometabolic risk factors. Sleep Med. 2014 Jan;15(1):42-50. doi: 10.1016/j.sleep.2013.09.012. Epub 2013 Oct 28. PMID 24333222
- [Background] Kroenke K, Strine TW, Spitzer RL, Williams JB, Berry JT, Mokdad AH. The PHQ-8 as a measure of current depression in the general population. J Affect Disord. 2009 Apr;114(1-3):163-73. doi: 10.1016/j.jad.2008.06.026. Epub 2008 Aug 27. PMID 18752852
- [Background] Knutson KL, Spiegel K, Penev P, Van Cauter E. The metabolic consequences of sleep deprivation. Sleep Med Rev. 2007 Jun;11(3):163-78. doi: 10.1016/j.smrv.2007.01.002. Epub 2007 Apr 17. PMID 17442599
- [Background] Morin CM, Belleville G, Belanger L, Ivers H. The Insomnia Severity Index: psychometric indicators to detect insomnia cases and evaluate treatment response. Sleep. 2011 May 1;34(5):601-8. doi: 10.1093/sleep/34.5.601. PMID 21532953
- [Background] Richey SM, Krystal AD. Pharmacological advances in the treatment of insomnia. Curr Pharm Des. 2011;17(15):1471-5. doi: 10.2174/138161211796197052. PMID 21476952
- [Background] Rusch HL, Rosario M, Levison LM, Olivera A, Livingston WS, Wu T, Gill JM. The effect of mindfulness meditation on sleep quality: a systematic review and meta-analysis of randomized controlled trials. Ann N Y Acad Sci. 2019 Jun;1445(1):5-16. doi: 10.1111/nyas.13996. Epub 2018 Dec 21. PMID 30575050
- [Background] Vyhlidal T, Dygryn J, Chmelik F. Actigraphy-Based Characteristics of Sleep in Paediatric Cancer Patients in Remission and a Comparison with Their Healthy Peers in the Recovery Stay. Nat Sci Sleep. 2022 Aug 25;14:1449-1456. doi: 10.2147/NSS.S374234. eCollection 2022. PMID 36045915
- [Derived] Staiano W, Callahan C, Davis M, Tanner L, Coe C, Kunkle S, Kirk U. Assessment of an App-Based Sleep Program to Improve Sleep Outcomes in a Clinical Insomnia Population: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2025 Apr 23;13:e68665. doi: 10.2196/68665. PMID 40267472